CLINICAL TRIAL: NCT06458179
Title: Retrospective Cohort Study for One Year Follow-up: Ultrasound Guided Radiofrequency Ablation of Proximal Greater Occipital Nerve is Effective
Brief Title: Ultrasound Guided Radiofrequency Ablation of Proximal Greater Occipital Nerve in Primary Occipital Neuralgia
Acronym: PGON-RFA
Status: Completed | Type: Observational
Sponsor: Mersin Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Suna Aşkın Turan, sponspor investigator, Mersin Training and Research Hospital
Other Study IDs: Occipital neuralgia
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Occipital Neuralgia
Keywords: headache; ultrasonography; greater occipital nerve; radiofrequency ablation
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Proximal greater occipital nerve radiofrequency ablation (RFA): Between January 1, 2022 and April 30, 2023, all patients diagnosed with primary unilateral occipital neuralgia who underwent US-guided diagnostic occipital nerve block and subsequent RFA of the PGON and were followed up for a minimum of one year were identified and included in the database. Patients lacking documentation or inadequate follow-up were excluded. Excluded from the study were patients with bilateral ON, secondary ON, other primary headaches, dermatitis or skin infections, and pacemakers. Based on clinical history and neurolgical examination (including Tinel's test), ON was diagnosed.
  Interventions: Procedure: Ultrasound-guided proximal greater occipital nerve radiofrequency ablation

INTERVENTIONS:
Procedure: Ultrasound-guided proximal greater occipital nerve radiofrequency ablation — In the prone position with the head slightly flexed and the US probe was placed in the neck transversely and then was located the bifid spinous process of C2 and the probe was lateralized (toward the affected side). At this level, the GON is located above the obliquus capitis inferior muscle and deeper than the semispinalis capitis muscle. The in-plane approach from medial to lateral was employed to treat the nerve with a 21 G 5-mm active tip radiofrequency needle. Sensory stimulation was administered at 50 Hz for 1 ms to induce paresthesia, pain, or irritation. A motor stimulus was applied at 2 Hz for 1 ms and up to 2 volts to see if fasciculation was absent. Then 1 mL of 2% lidocaine was administered through the RF cannulas to alleviate procedure related pain. Conventional RFA was conducted for 60 seconds at a temperature of 60 degrees. Following the procedure, 2 mg of dexamethasone was administered per lesion site.

SUMMARY:
The International Headache Society (IHS) defines occipital neuralgia, as a unilateral or bilateral paroxysmal, shooting, or stabbing pain in the posterior region of the scalp, in the distribution of the greater occipital nerve (GON), lesser occipital nerve (LON), or third occipital nerve (TON). The condition is occasionally accompanied by diminished sensation or dysesthesia in the affected area and is frequently associated with tenderness over the involved nerves. The majority of cases with occipital neuralgia are idiopathic, with no clearly defined anatomical cause. First, conservative treatment approaches including medication and physical therapy are frequently used. When conservative measures fail to alleviate occipital neuralgia, interventional treatments such as local occipital nerve anesthetic and corticosteroid infiltration, botulinum toxin A injection, occipital nerve subcutaneous neurostimulation or occipital nerve radifrequency treatment may be used.

DETAILED DESCRIPTION:
Radiofrequency ablation (RFA) is a thermal ablative procedure commonly used to treat chronic neurogenic pain by targeting peripheral nerves or dorsal root ganglion by destructing the tissue at a temperature ranging beteen 60-80 C. The pain is interrupted by destructing the nerve with Wallerian dejeneration. The pain interruption period is longer and stronger than pulsed radiofrequency. GON is a pure sensory nerve, RFA may be an alternative therapy option for occipital neuralgia. By ultrasound (US) guidance, at C2 level , GON lies between semispinalis capitis muscle and inferior oblique muscle. The GON is well identified here and can be easily targeted rather than trying to identify the terminal subcutaneous branches at the nuchal line. Diagnostic blockade was administered to patients who did not respond to conventional therapy. If the response to diagnostic blockade was greater than 50%, RFA was instituted one week later. Patients' headache intensity was measured using the Numeric Rating Scale-11 Pain Score (NRS) at each appointment (pre-intervention, 1-3-6, and 12 months post-intervention). At each appointment, an evaluation of headache disability was conducted using the Headache Impact Test (Hit-6) and the number of headache days per month. The efficacy of the treatment was defined as NRS<4 at the twelveth month. During the initial evaluation, patients' demographic details and headache symptoms were thoroughly questioned. In accordance with the Turkish National Headache and Pain Research Association's recommendation, patients were asked to keep up headache diaries for the duration of the treatment and all subsequent appointments. The headache intensity, headache disability and the number of headache days in a month, as well as the use of rescue medication, including NSAIDs and paracethamol, were determined from the diaries and discussed with the patient at each session.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral primary occipital neuralgia

Exclusion Criteria:

* Patients lacking documentation or inadequate follow-up
* Patients whom taking analgesic medication during the follow-up period
* Bilateral occipital neuralgia
* Secondary occipital neuralgia (e.g., cervical radiculopathy, infection, tumor, vascular compression of nerve, musculoskeletal diseases like C1-2 arthrosis)
* Other primary headaches
* Dermatitis or skin infections
* Pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients who underwent ultrasound-guided greater occipital nerve radiofrequency ablation for unilateal primary occipital neuralgia
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-04-29 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
NRS | Change from Baseline VAS at 1,3, 6 and 12 months
  Numerical rating scale (NRS) are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid (statistically measurable and reproducible) classification of symptom severity and disease control.

SECONDARY OUTCOMES:
Headache impact disability index (HIT-6) | Change from Baseline VAS at 1,3, 6 and 12 months
  These responses are summed to produce a total HIT-6 score that ranges from 36 to 78, where a higher score indicates a greater impact of headache on the daily life of the respondent. Scores can be interpreted using four groupings that indicate the severity of headache impact on the patient's life.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin Training and Research Hospital, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided